CLINICAL TRIAL: NCT01921920
Title: An Open-label, Randomized, Single-center, 4-way Crossover, Single Dose Bioequivalence Study Comparing Omeprazole 20 and 40-mg Aqueous Solvent Based Capsules Manufactured by AstraZeneca With Omeprazole 20 and 40-mg Organic-solvent Based Capsules Manufactured by Merck
Brief Title: Prilosec Bioequivalence Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D9584C00010
Record Dates: First submitted 2013-08-05; First posted 2013-08-14 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Bioequivalence, AUC, Cmax, Pharmacokinetics
Keywords: Omeprazole, Prilosec, Phase I, Healthy Subjects, Pharmacokinetics, Bioequivalence
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Omeprazole 20mg aqueous (Active Comparator): Treatment A: a single oral dose of omeprazole 20-mg aqueous-solvent based capsules (AstraZeneca - test)
  Interventions: Drug: Omeprazole
- Omeprazole 20mg organic (Active Comparator): Treatment B: a single oral dose of omeprazole 20-mg organic-solvent based capsules (Merck - reference for Treatment A)
  Interventions: Drug: Omeprazole
- Omeprazole 40mg aqueous (Active Comparator): Treatment C: a single dose of omeprazole 40-mg aqueous-solvent based capsules (AstraZeneca - test)
  Interventions: Drug: Omeprazole
- Omeprazole 40mg organic (Active Comparator): Treatment D: a single dose of omeprazole 40-mg organic-solvent based capsules (Merck - reference for Treatment C)
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Omeprazole 20 mg (AstraZeneca - test) Omeprazole 40 mg (AstraZeneca - test) Omeprazole 20 (Merck - reference) Omeprazole 40mg (Merck - reference)
  Other Names: Prilosec

SUMMARY:
This is An Open-label, Randomized, Single-center, 4-way Crossover, Single dose Bioequivalence Study Comparing Omeprazole 20 and 40-mg Aqueous solvent Based Capsules Manufactured by AstraZeneca with Omeprazole 20 and 40-mg Organic-solvent Based Capsules Manufactured by Merck

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18 to 50 years, inclusive, with suitable veins for cannulation or repeated venepuncture.
* Female could be of nonchildbearing potential (postmenopausal or irreversible surgical sterilization) and childbearing potential (negative pregnancy test at screening and use 2 effective methods of avoiding pregnancy).
* Have a body mass index (BMI) between 18 and 30 kg/m2, inclusive, and a weight of at least 50 kg and no more than 100 kg, inclusive.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in the physical examination, clinical laboratory values, 12-lead ECG, or vital signs, as judged by the Investigator.
* Moderate to heavy smokers (more than 10 cigarettes per day or equivalent in tobacco-containing products).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of omeprazole 20-mg aqueous-solvent based capsules versus omeprazole 20-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC
Bioequivalence of omeprazole 40-mg aqueous-solvent based capsules versus omeprazole 40-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC
Bioequivalence of omeprazole 20-mg aqueous-solvent based capsules versus omeprazole 20-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC (0-t)
Bioequivalence of omeprazole 20-mg aqueous-solvent based capsules versus omeprazole 20-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  Cmax
Bioequivalence of omeprazole 40-mg aqueous-solvent based capsules versus omeprazole 40-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC(0-t)
Bioequivalence of omeprazole 40-mg aqueous-solvent based capsules versus omeprazole 40-mg organic solvent based capsules | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  Cmax

SECONDARY OUTCOMES:
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  Cmax
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  Cmax
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  t1/2
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  tmax
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC(0-t)
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 20-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  λz
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  tmax
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC(0-t)
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  AUC
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  λz
Pharmacokinetics of 2 enteric-coated formulations after a single dose of 40-mg omeprazole | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours postdose.
  t1/2

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles Phase I unit, Kansas; Helen Lunde, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States